CLINICAL TRIAL: NCT03592914
Title: Respiratory Rate Accuracy Verification Clinical: Pulmonary Rehabilitation
Brief Title: Respiratory Rate Accuracy Verification Clinical: Pulmonary Rehabilitation Patients
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Collaborators: Valley Inspired Products (Unknown)
Responsible Party: Sponsor
Other Study IDs: QATP3161
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subjects with respiratory disease: This study is a comparative, single-center study. This is a minimal risk study using a non-significant risk device. A minimum of 60 and maximum of 70 subjects will be enrolled in the study. Subject participation will last approximately 1 hour(s).

SUMMARY:
Study Design: This study is a comparative, single-center study. This is a minimal risk study (as defined in 21 CFR Part 56) using a non-significant risk device (as defined in 21 CFR Part 812.3). A minimum of 60 subjects will be enrolled in the study. Subject participation will last approximately 1 hour.

DETAILED DESCRIPTION:
Study Design: This study is a comparative, single-center study. This is a minimal risk study (as defined in 21 CFR Part 56) using a non-significant risk device (as defined in 21 CFR Part 812.3). A minimum of 60 subjects will be enrolled in the study. Subject participation will last approximately 1 hour.

Objective(s):

The primary objective of this study is to evaluate the two Fingertip Respiratory Rate (FTRR) algorithms performance of Nonin's Onyx 3 by attempting to demonstrate a mean error for FTRR < 1.0 BPM during spontaneous breathing.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years old;
* The subject has given written informed consent to participate in the study;
* The subject is both willing and able to comply with study procedures.

Exclusion Criteria:

* The subject has a history of or current atrial fibrillation;
* The subject has a documented history of frequent premature ventricular contractions (PVCs), defined as >3 per 30 seconds;
* The subject has an implanted pacemaker;
* The subject has had any relevant injury at the sensor location site (self-reported);
* The subject has deformities or abnormalities that may prevent proper application of the device under test (based on examination);
* The subject is currently or trying to get pregnant (self-reported); and/or
* The subject has another health condition which in the opinion of the principal investigator makes subject unsuitable for testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who might be seen in a respiratory rehabilitation center.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Evaluate the two Fingertip Respiratory Rate (FTRR) algorithms performance of Nonin's Onyx 3 | 40 minutes
  Measure respiratory rates

CONTACTS AND LOCATIONS:
Locations (1):
- Nonin Medical, Inc., Plymouth, Minnesota, United States